CLINICAL TRIAL: NCT05062486
Title: An Open-Label, Randomized, Double Arm, Phase 2 Study to Evaluate the Safety and Efficacy of C and RQC for Preventing Progression in Age-Related Macular Degeneration
Brief Title: A Study to Evaluate the Safety and Efficacy of RQC for AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paul A Knepper, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Paul A Knepper, MD PhD, Sponsor-Investigator, Zaparackas and Knepper LTD
Organization: Zaparackas and Knepper LTD (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZK-01-2021
Record Dates: First submitted 2021-09-08; First posted 2021-09-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Age-related Macular Degeneration
Keywords: Curcumin; Resveratrol; Quercetin; Macular Degeneration, Age-Related; Age-Related Maculopathy; Adult Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Resveratrol; Quercetin; Curcumin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resveratrol, Quercetin, Curcumin (RQC) (Experimental): Resveratrol (100mg BID), Quercetin (120mg BID), Curcumin (1000mg BID); 24 months
  Interventions: Drug: Resveratrol, Quercetin, Curcumin (RQC)
- Curcumin (Active Comparator): Curcumin (1000mg BID); 24 months
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Resveratrol, Quercetin, Curcumin (RQC) — 100 mg resveratrol, 120 mg quercetin, 1000 mg curcumin BID
  Arms: Resveratrol, Quercetin, Curcumin (RQC)
Drug: Curcumin — 1000 mg curcumin BID
  Arms: Curcumin

SUMMARY:
To evaluate the safety and efficacy of resveratrol, quercetin, and curcumin in combination (RQC) over 2 years in patients with age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
The objective of the study is to institute an open-label, randomized, double arm, phase 2 study to evaluate the safety and efficacy of resveratrol, quercetin, and curcumin in combination (RQC) versus curcumin alone (C) in AMD. The primary outcomes are change in drusen volume, geographic atrophy growth rate, and progression to moderate vision loss. Progression to advanced AMD will serve as a secondary outcome measure. Participants are classified by pre-AMD severity at baseline and randomized into either the C (n=50) or RQC (n=150) arm. Curcumin is taken orally at a dose of 1000 mg twice per day. RQC is taken orally at a dose of 100 mg resveratrol, 120 mg quercetin, and 1000 mg curcumin twice per day. The study will be conducted over 2 years with follow-up visits at least every 6 months.

Safety is evaluated using adverse event reporting, vital sign/physical examinations, and blood testing. Efficacy is evaluated using a series of OCT-based retinal photography and image processing techniques to measure drusen volume, GA area, and the presence of advanced disease (GA or wet AMD). Progression to moderate vision loss is defined as a loss of 15 letters on the Early Treatment for Diabetic Retinopathy Study (ETDRS) charts. The status of 15 single nucleotide polymorphisms reported to be associated with AMD are analyzed and incorporated as covariates into multivariate models of primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race or ethnicity.
2. Aged 50-90 years at time of study entry.
3. Ability to speak, read, and understand English.
4. Ability to take oral medication and be willing to adhere to the study regimen.
5. Capable of providing informed consent/provision of signed and dated informed consent.
6. Stated willingness to comply with all procedures and availability for the duration of the study.
7. Diagnosis of dry AMD (AREDS categories Early, drusen 63-124 µm in width; Intermediate, drusen ≥125 µm in width; or Advanced, macular geographic atrophy) as documented by OCT and/or color retinal photography.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 90 days.
2. The presence of wet AMD.
3. The presence of ocular disease or condition that may confound evaluation of the retina or could require medical or surgical intervention.
4. Previous retinal or other ocular surgical procedures (other than cataract extraction) that may have complicated assessment of the progression of AMD.
5. A serious or complex systemic medical disease or condition with a poor five-year survival prognosis or that would make adherence or follow-up difficult or unlikely.
6. Diagnosis of Alzheimer's disease or dementia, diagnosis of a serious gastrointestinal or stomach condition, or positive for HIV, hepatitis B surface antigen, or hepatitis C antibodies.
7. History of inherited bleeding disorder.
8. Use of any anticoagulant medication within 5 days before the first dose of investigative product is scheduled or required for subsequent medical treatment in the course of the study.
9. Clinically significant abnormal physical examination/vital signs or laboratory and coagulation blood tests as deemed appropriate by the investigator.
10. History of or a reason to believe participant has a history of drug or alcohol abuse within the past 5 years.
11. History of known allergy to any component of the investigational product.
12. Preplanned surgery or procedures that would interfere with the conduct of the study.
13. Currently incarcerated prisoners.
14. Currently pregnant or lactating.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Change in Drusen Volume from Baseline | 24 months
  Macular drusen volume measured in µm3.
Geographic Atrophy (GA) Growth Rate | 24 months
  The annual growth rate of GA or nascent GA area measured in mm2.
Progression to Moderate Vision Loss | 24 months
  Progression defined as a decrease in ETDRS BCVA score of 15 or more letters.
Adverse Events | 24 months
  Safety outcomes include adverse and serious adverse events and vital sign/physical examination tests.

SECONDARY OUTCOMES:
Progression to Advanced AMD | 24 months
  Progression defined as the development of geographic atrophy or choroidal neovascularization detected by OCT imaging using autofluorescence, infrared, and/or angiography modules.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Knepper, MD, PhD, Principal Investigator — Zaparackas Knepper, Ltd; Zibute Zaparackas, MD, Principal Investigator — Zaparackas Knepper, Ltd
Locations (1):
- Zaparackas M.D. & Knepper M.D. Ph.D., Ltd, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almeida L, Vaz-da-Silva M, Falcao A, Soares E, Costa R, Loureiro AI, Fernandes-Lopes C, Rocha JF, Nunes T, Wright L, Soares-da-Silva P. Pharmacokinetic and safety profile of trans-resveratrol in a rising multiple-dose study in healthy volunteers. Mol Nutr Food Res. 2009 May;53 Suppl 1:S7-15. doi: 10.1002/mnfr.200800177. PMID 19194969
- [Background] Ambati J, Fowler BJ. Mechanisms of age-related macular degeneration. Neuron. 2012 Jul 12;75(1):26-39. doi: 10.1016/j.neuron.2012.06.018. PMID 22794258
- [Background] Barratt-Due A, Pischke SE, Nilsson PH, Espevik T, Mollnes TE. Dual inhibition of complement and Toll-like receptors as a novel approach to treat inflammatory diseases-C3 or C5 emerge together with CD14 as promising targets. J Leukoc Biol. 2017 Jan;101(1):193-204. doi: 10.1189/jlb.3VMR0316-132R. Epub 2016 Aug 31. PMID 27581539
- [Background] Boocock DJ, Faust GE, Patel KR, Schinas AM, Brown VA, Ducharme MP, Booth TD, Crowell JA, Perloff M, Gescher AJ, Steward WP, Brenner DE. Phase I dose escalation pharmacokinetic study in healthy volunteers of resveratrol, a potential cancer chemopreventive agent. Cancer Epidemiol Biomarkers Prev. 2007 Jun;16(6):1246-52. doi: 10.1158/1055-9965.EPI-07-0022. PMID 17548692
- [Background] Brown VA, Patel KR, Viskaduraki M, Crowell JA, Perloff M, Booth TD, Vasilinin G, Sen A, Schinas AM, Piccirilli G, Brown K, Steward WP, Gescher AJ, Brenner DE. Repeat dose study of the cancer chemopreventive agent resveratrol in healthy volunteers: safety, pharmacokinetics, and effect on the insulin-like growth factor axis. Cancer Res. 2010 Nov 15;70(22):9003-11. doi: 10.1158/0008-5472.CAN-10-2364. Epub 2010 Oct 8. PMID 20935227
- [Background] Byun EB, Yang MS, Choi HG, Sung NY, Song DS, Sin SJ, Byun EH. Quercetin negatively regulates TLR4 signaling induced by lipopolysaccharide through Tollip expression. Biochem Biophys Res Commun. 2013 Feb 22;431(4):698-705. doi: 10.1016/j.bbrc.2013.01.056. Epub 2013 Jan 24. PMID 23353651
- [Background] Chainani-Wu N. Safety and anti-inflammatory activity of curcumin: a component of tumeric (Curcuma longa). J Altern Complement Med. 2003 Feb;9(1):161-8. doi: 10.1089/107555303321223035. PMID 12676044
- [Background] Cheng AL, Hsu CH, Lin JK, Hsu MM, Ho YF, Shen TS, Ko JY, Lin JT, Lin BR, Ming-Shiang W, Yu HS, Jee SH, Chen GS, Chen TM, Chen CA, Lai MK, Pu YS, Pan MH, Wang YJ, Tsai CC, Hsieh CY. Phase I clinical trial of curcumin, a chemopreventive agent, in patients with high-risk or pre-malignant lesions. Anticancer Res. 2001 Jul-Aug;21(4B):2895-900. PMID 11712783
- [Background] AREDS2 Research Group; Chew EY, Clemons T, SanGiovanni JP, Danis R, Domalpally A, McBee W, Sperduto R, Ferris FL. The Age-Related Eye Disease Study 2 (AREDS2): study design and baseline characteristics (AREDS2 report number 1). Ophthalmology. 2012 Nov;119(11):2282-9. doi: 10.1016/j.ophtha.2012.05.027. Epub 2012 Jul 26. PMID 22840421
- [Background] Chew EY, Lindblad AS, Clemons T; Age-Related Eye Disease Study Research Group. Summary results and recommendations from the age-related eye disease study. Arch Ophthalmol. 2009 Dec;127(12):1678-9. doi: 10.1001/archophthalmol.2009.312. No abstract available. PMID 20008727
- [Background] Cottart CH, Nivet-Antoine V, Beaudeux JL. Review of recent data on the metabolism, biological effects, and toxicity of resveratrol in humans. Mol Nutr Food Res. 2014 Jan;58(1):7-21. doi: 10.1002/mnfr.201200589. Epub 2013 Jun 6. PMID 23740855
- [Background] Davis MD, Gangnon RE, Lee LY, Hubbard LD, Klein BE, Klein R, Ferris FL, Bressler SB, Milton RC; Age-Related Eye Disease Study Group. The Age-Related Eye Disease Study severity scale for age-related macular degeneration: AREDS Report No. 17. Arch Ophthalmol. 2005 Nov;123(11):1484-98. doi: 10.1001/archopht.123.11.1484. PMID 16286610
- [Background] Dhillon N, Aggarwal BB, Newman RA, Wolff RA, Kunnumakkara AB, Abbruzzese JL, Ng CS, Badmaev V, Kurzrock R. Phase II trial of curcumin in patients with advanced pancreatic cancer. Clin Cancer Res. 2008 Jul 15;14(14):4491-9. doi: 10.1158/1078-0432.CCR-08-0024. PMID 18628464
- [Background] Egert S, Wolffram S, Bosy-Westphal A, Boesch-Saadatmandi C, Wagner AE, Frank J, Rimbach G, Mueller MJ. Daily quercetin supplementation dose-dependently increases plasma quercetin concentrations in healthy humans. J Nutr. 2008 Sep;138(9):1615-21. doi: 10.1093/jn/138.9.1615. PMID 18716159
- [Background] Ferris FL 3rd, Bailey I. Standardizing the measurement of visual acuity for clinical research studies: Guidelines from the Eye Care Technology Forum. Ophthalmology. 1996 Jan;103(1):181-2. doi: 10.1016/s0161-6420(96)30742-2. No abstract available. PMID 8628551
- [Background] Ferris FL 3rd, Wilkinson CP, Bird A, Chakravarthy U, Chew E, Csaky K, Sadda SR; Beckman Initiative for Macular Research Classification Committee. Clinical classification of age-related macular degeneration. Ophthalmology. 2013 Apr;120(4):844-51. doi: 10.1016/j.ophtha.2012.10.036. Epub 2013 Jan 16. PMID 23332590
- [Background] Ferry DR, Smith A, Malkhandi J, Fyfe DW, deTakats PG, Anderson D, Baker J, Kerr DJ. Phase I clinical trial of the flavonoid quercetin: pharmacokinetics and evidence for in vivo tyrosine kinase inhibition. Clin Cancer Res. 1996 Apr;2(4):659-68. PMID 9816216
- [Background] Feuer WJ, Yehoshua Z, Gregori G, Penha FM, Chew EY, Ferris FL, Clemons TE, Lindblad AS, Rosenfeld PJ. Square root transformation of geographic atrophy area measurements to eliminate dependence of growth rates on baseline lesion measurements: a reanalysis of age-related eye disease study report no. 26. JAMA Ophthalmol. 2013 Jan;131(1):110-1. doi: 10.1001/jamaophthalmol.2013.572. No abstract available. PMID 23307222
- [Background] Gradisar H, Keber MM, Pristovsek P, Jerala R. MD-2 as the target of curcumin in the inhibition of response to LPS. J Leukoc Biol. 2007 Oct;82(4):968-74. doi: 10.1189/jlb.1206727. Epub 2007 Jul 3. PMID 17609337
- [Background] Grunwald JE, Pistilli M, Ying GS, Maguire MG, Daniel E, Martin DF; Comparison of Age-related Macular Degeneration Treatments Trials Research Group. Growth of geographic atrophy in the comparison of age-related macular degeneration treatments trials. Ophthalmology. 2015 Apr;122(4):809-16. doi: 10.1016/j.ophtha.2014.11.007. Epub 2014 Dec 24. PMID 25542520
- [Background] Gupta SC, Patchva S, Aggarwal BB. Therapeutic roles of curcumin: lessons learned from clinical trials. AAPS J. 2013 Jan;15(1):195-218. doi: 10.1208/s12248-012-9432-8. Epub 2012 Nov 10. PMID 23143785
- [Background] Handa JT, Bowes Rickman C, Dick AD, Gorin MB, Miller JW, Toth CA, Ueffing M, Zarbin M, Farrer LA. A systems biology approach towards understanding and treating non-neovascular age-related macular degeneration. Nat Commun. 2019 Jul 26;10(1):3347. doi: 10.1038/s41467-019-11262-1. PMID 31350409
- [Background] Hewlings SJ, Kalman DS. Curcumin: A Review of Its Effects on Human Health. Foods. 2017 Oct 22;6(10):92. doi: 10.3390/foods6100092. PMID 29065496
- [Background] Jobin C, Bradham CA, Russo MP, Juma B, Narula AS, Brenner DA, Sartor RB. Curcumin blocks cytokine-mediated NF-kappa B activation and proinflammatory gene expression by inhibiting inhibitory factor I-kappa B kinase activity. J Immunol. 1999 Sep 15;163(6):3474-83. PMID 10477620
- [Background] Keenan TD, Agron E, Domalpally A, Clemons TE, van Asten F, Wong WT, Danis RG, Sadda S, Rosenfeld PJ, Klein ML, Ratnapriya R, Swaroop A, Ferris FL 3rd, Chew EY; AREDS2 Research Group. Progression of Geographic Atrophy in Age-related Macular Degeneration: AREDS2 Report Number 16. Ophthalmology. 2018 Dec;125(12):1913-1928. doi: 10.1016/j.ophtha.2018.05.028. Epub 2018 Jul 27. PMID 30060980
- [Background] la Porte C, Voduc N, Zhang G, Seguin I, Tardiff D, Singhal N, Cameron DW. Steady-State pharmacokinetics and tolerability of trans-resveratrol 2000 mg twice daily with food, quercetin and alcohol (ethanol) in healthy human subjects. Clin Pharmacokinet. 2010 Jul;49(7):449-54. doi: 10.2165/11531820-000000000-00000. PMID 20528005
- [Background] Merle NS, Paule R, Leon J, Daugan M, Robe-Rybkine T, Poillerat V, Torset C, Fremeaux-Bacchi V, Dimitrov JD, Roumenina LT. P-selectin drives complement attack on endothelium during intravascular hemolysis in TLR-4/heme-dependent manner. Proc Natl Acad Sci U S A. 2019 Mar 26;116(13):6280-6285. doi: 10.1073/pnas.1814797116. Epub 2019 Mar 8. PMID 30850533
- [Background] Pennington KL, DeAngelis MM. Epidemiology of age-related macular degeneration (AMD): associations with cardiovascular disease phenotypes and lipid factors. Eye Vis (Lond). 2016 Dec 22;3:34. doi: 10.1186/s40662-016-0063-5. eCollection 2016. PMID 28032115
- [Background] Seddon JM, Silver RE, Kwong M, Rosner B. Risk Prediction for Progression of Macular Degeneration: 10 Common and Rare Genetic Variants, Demographic, Environmental, and Macular Covariates. Invest Ophthalmol Vis Sci. 2015 Apr;56(4):2192-202. doi: 10.1167/iovs.14-15841. PMID 25655794
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Vadhan-Raj S, Weber DM, Wang M, Giralt SA, Thomas SK, Alexanian R, Zhou X, Patel P, Bueso-Ramos CE, Newman RA, Aggarwal BB. Curcumin downregulates NF-kB and related genes in patients with multiple myeloma: results of a phase I/II study. Blood. 2007;110(11):1177.
- [Background] Wong WL, Su X, Li X, Cheung CM, Klein R, Cheng CY, Wong TY. Global prevalence of age-related macular degeneration and disease burden projection for 2020 and 2040: a systematic review and meta-analysis. Lancet Glob Health. 2014 Feb;2(2):e106-16. doi: 10.1016/S2214-109X(13)70145-1. Epub 2014 Jan 3. PMID 25104651
- [Background] Youn HS, Lee JY, Fitzgerald KA, Young HA, Akira S, Hwang DH. Specific inhibition of MyD88-independent signaling pathways of TLR3 and TLR4 by resveratrol: molecular targets are TBK1 and RIP1 in TRIF complex. J Immunol. 2005 Sep 1;175(5):3339-46. doi: 10.4049/jimmunol.175.5.3339. PMID 16116226
- [Background] Youn HS, Saitoh SI, Miyake K, Hwang DH. Inhibition of homodimerization of Toll-like receptor 4 by curcumin. Biochem Pharmacol. 2006 Jun 28;72(1):62-9. doi: 10.1016/j.bcp.2006.03.022. Epub 2006 Apr 1. PMID 16678799
- [Background] Koronyo Y, Biggs D, Barron E, Boyer DS, Pearlman JA, Au WJ, Kile SJ, Blanco A, Fuchs DT, Ashfaq A, Frautschy S, Cole GM, Miller CA, Hinton DR, Verdooner SR, Black KL, Koronyo-Hamaoui M. Retinal amyloid pathology and proof-of-concept imaging trial in Alzheimer's disease. JCI Insight. 2017 Aug 17;2(16):e93621. doi: 10.1172/jci.insight.93621. eCollection 2017 Aug 17. PMID 28814675
- [Background] Koronyo-Hamaoui M, Koronyo Y, Ljubimov AV, Miller CA, Ko MK, Black KL, Schwartz M, Farkas DL. Identification of amyloid plaques in retinas from Alzheimer's patients and noninvasive in vivo optical imaging of retinal plaques in a mouse model. Neuroimage. 2011 Jan;54 Suppl 1:S204-17. doi: 10.1016/j.neuroimage.2010.06.020. Epub 2010 Jun 13. PMID 20550967